CLINICAL TRIAL: NCT06388278
Title: Cost-effectiveness Analysis of an Antimicrobial Stewardship Program in Regione Lombardia: "Finalizzata di Rete 2018"
Brief Title: Cost-effectiveness Analysis of an Antimicrobial Stewardship Program in Regione Lombardia (RF-net2018)
Acronym: RF-net2018
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Regione Lombardia (Other); Ministero della Salute, Italy (Other)
Responsible Party: Principal Investigator, malattie_infettive, Alessandra Bandera, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: NET-2018-12366982-4/ASP_LOMB
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Antimicrobial Stewardship; Cost-effectiveness Analysis
Keywords: antimicrobial stewardship; cost-effectiveness analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cost-effectiveness analysis of an Antimicrobial Stewardship program in Regione Lombardia: "RF-net2018" is a prospective, experimental, multicenter, pre-post study, whose objectives are the evaluation of the efficiency of economic resources allocated to the antimicrobial stewardship program (AMS) in patients with infection and in patients with infections caused by carbapenem-resistant gram-negative (CR-GN) bacteria, identified in a network of 18 hospital facilities participating in our study. Moreover, this study aims to compare hospital mortality among patients admitted to the facilities participating in the study before and during the implementation of the AMS project. The study will include two main phases of analysis: the pre-intervention-phase and the intervention phase, both of 6 months duration. The pre-intervention phase will serve as a control for the intervention phase. The intervention phase is represented by antimicrobial stewardship activities which have been implemented in the network of 18 hospital facilities and that include a group of activities listed above (Hospital commitment, Tracking and reporting, Action and Education). Data source and analysis for the cost-effectiveness analysis, using month-department as statistical unit, are regional data: Discharge record ICD-9 codes (identification of target population 1, 2, 3, average days of hospitalization and mortality), R file (for antibiotic drug consumption month-ward) and Microbio (identification of target population 2, CR-GN and MRSA bacteremia and Cases of C. difficile infection). For what concerns healthcare costs data, each Management control office of the 18 facilities has to provide: AVERAGE HOSPITALISATION DAYS, NUMBER OF HOSPITALIZED AND TRANSFERRED PATIENTS and HEALTHCARE COSTS (healthcare personnel, diagnostic services, surgical interventions and consumption of operating rooms).

DETAILED DESCRIPTION:
Cost-effectiveness analysis of an Antimicrobial Stewardship program in Regione Lombardia: "Finalizzata di Rete 2018" is a prospective, experimental, multicenter, pre-post study. The objectives of this study are:

* Objective 1: evaluate the efficiency of the economic resources allocated to the antimicrobial stewardship program (AMS) through a cost-effectiveness analysis in patients with infection. These patients will be identified in a network of 18 hospital facilities participating in our study
* Objective 2: evaluate the efficiency of the economic resources allocated to the AMS program through a cost-effectiveness analysis in patients with infections caused by carbapenem-resistant gram-negative (CR-GN) bacteria. These patients will be identified in a network of 18 hospital facilities participating in our study
* Objective 3: compare hospital mortality among patients admitted to the facilities participating in the study before and during the implementation of the AMS project

Study population for different objectives are:

* For Objective 1 and 3: All hospitalizations of subjects aged 18 years or older whose Hospital Discharge Form (SDO) contains at least one ICD-9-CM code that belongs to the list of codes that identify hospitalizations that likely included the administration of antimicrobial therapy (ongoing consensus activity)
* For Objective 2: Subgroup of the population included for objectives 1 and 3 in which bacteremia due to carbapenem-resistant bacteria has been identified

The study will include two main phases of analysis:

* The pre-intervention-phase (6 months)
* The intervention-phase (6 months)

The pre-intervention phase will serve as a control for the intervention phase and the unit of measurement used is month-department

Intervention phase is represented by antimicrobial stewardship activities which have been implemented in the network of 18 hospital facilities and that include:

⦁ HOSPITAL COMMITMENT : A. Definition of an official group of specialists responsible for antimicrobial stewardship activities (infectious diseases specialist, IPC referent, pharmacist e microbiologist).

B. Presence of a multidisciplinary reference team that includes representatives from other medical specialties (in addition to the figures reported in point A.)

⦁ TRACKING AND REPORTING A. Monitoring the quality/adequacy of antimicrobial use at the unit and/or hospital level by hospital management B. Control of the quantity of antimicrobials prescribed/dispensed/purchased at unit level and/or hospital level by hospital management C. Monthly/bimonthly/quarterly/half-yearly report of antibiotic consumption for each department with circulation of these reports at intra-hospital level.

D. Monthly/bimonthly/quarterly/semiannual reporting of cases of C. difficile infection, carbapenem-resistant gram negative bacteria isolated from blood cultures and methicillin-resistant S.aureus (MRSA) with subsequent circulation of these reports at intra-hospital level.

* ACTION A. Infectious disease review of carbapenem prescription (in any form) B. Ward rounds focusing on infection management or antibiotic prescribing in departments in your hospital
* EDUCATION A. Training events aimed at medical and nursing healthcare personnel with a focus on the use of antibiotics belonging to the carbapenem family and on controlling the spread of multidrug-resistant (MDR) microorganisms

ELIGIBILITY:
Inclusion Criteria:

* All hospitalizations of subjects aged 18 years or older whose Hospital Discharge Form (SDO) contains at least one ICD-9-CM code that belongs to the list of codes that identify hospitalizations that likely included the administration of antimicrobial therapy
* Subgroup of the population included for objectives 1 and 3 in which bacteremia due to carbapenem-resistant bacteria has been identified

Exclusion Criteria:

* patients non included in Inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population for different objectives are:
  * For Objective 1 and 3: All hospitalizations of subjects aged 18 years or older whose Hospital Discharge Form (SDO) contains at least one ICD-9-CM code that belongs to the list of codes that identify hospitalizations that likely included the administration of antimicrobial therapy (ongoing consensus activity)
  * For Objective 2: Subgroup of the population included for objectives 1 and 3 in which bacteremia due to carbapenem-resistant bacteria has been identified
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
evaluate the efficiency of the economic resources allocated to the antimicrobial stewardship program (AMS) through a cost-effectiveness analysis in patients with infection | 12 months
  evaluate the efficiency of the economic resources allocated to the antimicrobial stewardship program (AMS) through a cost-effectiveness analysis in patients with infection. These patients will be identified in a network of 18 hospital facilities participating in our study
evaluate the efficiency of the economic resources allocated to the AMS program through a cost-effectiveness analysis in patients with infections caused by carbapenem-resistant gram-negative (CR-GN) bacteria. | 12 months
  evaluate the efficiency of the economic resources allocated to the AMS program through a cost-effectiveness analysis in patients with infections caused by carbapenem-resistant gram-negative (CR-GN) bacteria. These patients will be identified in a network of 18 hospital facilities participating in our study
compare hospital mortality among patients admitted to the facilities participating in the study before and during the implementation of the AMS project | 12 months
  compare hospital mortality among patients admitted to the facilities participating in the study before and during the implementation of the AMS project. These patients will be identified in a network of 18 hospital facilities participating in our study

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Gori, Principal Investigator — IRCCS Fondazione Cà Granda Policlinico of Milan
Locations (1):
- IRCCS Fondazione Policlinico of Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided